CLINICAL TRIAL: NCT03363841
Title: Open-Label Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of Oral Ibrexafungerp (SCY-078) as an Emergency Use Treatment for Patients With Candidiasis, Including Candidemia, Caused by Candida Auris
Brief Title: Open-Label Study to Evaluate the Efficacy and Safety of Oral Ibrexafungerp (SCY-078) in Patients With Candidiasis Caused by Candida Auris (CARES)
Acronym: CARES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scynexis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCY-078-305
Record Dates: First submitted 2017-11-14; First posted 2017-12-06 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Candidiasis, Invasive; Candidemia
Keywords: Candida auris
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia | interventions — ibrexafungerp

STUDY DESIGN:
Intervention Model Description: non comparator, single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SCY-078 (Experimental): SCY-078
  Interventions: Drug: SCY-078

INTERVENTIONS:
Drug: SCY-078 — Oral SCY-078

SUMMARY:
This is a multicenter, open-label, non-comparator, single-arm study to evaluate the efficacy, safety, tolerability and PK (pharmacokinetics) of oral SCY-078 as an emergency use treatment for patients with a documented Candida auris infection.

DETAILED DESCRIPTION:
This is a multicenter, open-label, non-comparator, single-arm study to evaluate the efficacy, safety, tolerability and PK (for a subset of subjects) of oral SCY-078 in male and female subjects ≥18 years of age with a documented Candida auris infection. Patients will be treated with SCY-078 for up to 90 days.

Subjects must have a documented candidiasis, including candidemia, caused by Candida auris to be considered for enrollment. Subjects are also eligible if they are receiving intravenous (IV) antifungal therapy for their C. auris infection and, in the judgment of the investigator, continued IV antifungal therapy is not feasible or desirable due to clinical or logistical circumstances. Subjects must meet all study criteria to be eligible for inclusion. Inclusion of each subject in the study must be approved by the Sponsor prior to enrollment.

Following a screening visit , there will be up to 11 treatment visits, a follow-up visit and 2 follow-up contacts (survival visits)

ELIGIBILITY:
Inclusion Criteria:

* Subject must fulfill the following KEY criteria to be eligible for study admission:

  1. Subject is a male or female adult ≥ 18 years of age on the day the study informed consent form (ICF) is signed.
  2. Subject has a documented candidiasis, including candidemia, caused by Candida auris. The subject is also eligible if he/she is receiving IV antifungal therapy for their C. auris infection and, in the judgment of the investigator, long-term IV antifungal therapy is not feasible or desirable due to clinical or logistical circumstances. A documented candidiasis, including candidemia, caused by Candida auris is defined as the recovery of Candida auris by culture of a sample obtained within the last 7 days.
  3. Subject is able to tolerate medication orally or through a nasogastric (NG) tube or percutaneous endoscopic gastrostomy (PEG) tube.

Exclusion Criteria:

* KEY exclusion criteria:

  1. Subject has a fungal disease with central nervous system involvement.
  2. Subject has a fungal disease of the bone and/or joint that is expected to require >90 days of study drug treatment.
  3. Subject has an inappropriately controlled fungal infection source (e.g., persistent catheters, devices, identified abscess) that is likely the source of the fungal infection.
  4. Subject is hemodynamically unstable and/or requiring vasopressor medication for blood pressure support.
  5. Subject has abnormal liver test parameters: AST or ALT >10 x ULN, and/or total bilirubin >5 x ULN. Note: Subjects with unconjugated hyperbilirubinemia with diagnosis of Gilbert's disease are not excluded.
  6. Subject has an Apache score >16.
  7. Subject has serum creatinine >3 times from Baseline (Screening/Treatment Day 1) value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Angulo, MD, Study Director — Scynexis, Inc.
Locations (12):
- Scynexis, Inc., Jersey City, New Jersey, United States
- India (5):
  - St John's Medical College and Hospital, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences (AIMS), Kanayannur, Kochi
  - Institute of Critical Care Medicine Max Super Specialty Hospital, Saket, New Delhi
  - King George Medical University, Lucknow, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research, Department of Anaesthesia and special care, Chandigarh
- Aga Khan University Hospital, Karachi, Sindh, Pakistan
- South Africa (5):
  - Johese Clinical Research, Unitas Hospital Centurion,, South Africa, 0157, Centurion, Gauteng
  - Emmed Research, Jakarta Hospital, Pretoria, Gauteng
  - Into Research, Life Groenkloof Hospital, Pretoria, Gauteng
  - Johese Clinical Research, Midstream, Pretoria, Gauteng
  - Zuid Afrikaans Hospital, Pretoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Berkow EL, Angulo D, Lockhart SR. In Vitro Activity of a Novel Glucan Synthase Inhibitor, SCY-078, against Clinical Isolates of Candida auris. Antimicrob Agents Chemother. 2017 Jun 27;61(7):e00435-17. doi: 10.1128/AAC.00435-17. Print 2017 Jul. No abstract available. PMID 28483955
- [Background] Larkin E, Hager C, Chandra J, Mukherjee PK, Retuerto M, Salem I, Long L, Isham N, Kovanda L, Borroto-Esoda K, Wring S, Angulo D, Ghannoum M. The Emerging Pathogen Candida auris: Growth Phenotype, Virulence Factors, Activity of Antifungals, and Effect of SCY-078, a Novel Glucan Synthesis Inhibitor, on Growth Morphology and Biofilm Formation. Antimicrob Agents Chemother. 2017 Apr 24;61(5):e02396-16. doi: 10.1128/AAC.02396-16. Print 2017 May. PMID 28223375

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 34 Participants Screened, 30 met the selection criteria for the study
Period: Overall Study
Arm/Group | SCY-078
Started | 30
Completed | 20
Not Completed | 10
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Death | 7
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Ibrexafungerp 750 mg: Oral ibrexafungerp was to be given as 750 mg BID (total daily dose = 1500 mg) on Days 1 and 2, followed by oral ibrexafungerp 750 mg QD (total daily dose = 750 mg) from Day 3 onwards for up to 90 days
Arm/Group | Ibrexafungerp 750 mg
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 60.3 [23.0 to 97.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Global Success at End of Treatment as Determined by the Data Monitoring Committee
Description: The percentage of participants with global success at End of Treatment (EoT) as determined by the Data Monitoring Committee. Global success is defined as complete or partial resolution of signs and symptoms associated with the fungal disease and mycological eradication.
Time Frame: At (EoT) Visit (up to 90 days after Day 1)
Population: Intent to Treat Population (ITT): all subjects who were enrolled in the study
Measure: Count of Participants; unit: Participants
Groups:
- Ibrexafungerp 750mg: Oral ibrexafungerp was to be given as 750 mg BID (total daily dose = 1500 mg) on Days 1 and 2, followed by oral ibrexafungerp 750 mg QD (total daily dose = 750 mg) from Day 3 onwards for up to 90 days
Arm/Group | Ibrexafungerp 750mg
Number analyzed (Participants) | 30
Participants | 21

2. Secondary Outcome: Percent of Participants With Treatment-emergent Adverse Events
Description: Percent of participants with treatment-emergent Adverse Events (TEAEs)
Time Frame: Through study completion, up to 132 days
Population: Safety Population: any participant that received at least one dose of study medication and had at least one safety assessment post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 750 mg
Number analyzed (Participants) | 30
Participants | 25

3. Secondary Outcome: Number of Participants Discontinued Due to Adverse Events
Description: Number of participants with Discontinuations due to Adverse Events
Time Frame: Through study completion (up to 132 Days)
Population: Safety Population - any participant that received at least one dose of study medication and had at least one safety assessment post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 750 mg
Number analyzed (Participants) | 30
Participants | 1

4. Secondary Outcome: Percentage of Participants With Recurrence of Baseline Fungal Infection
Description: The percentage of participants with a recurrence of the baseline fungal infection at the 6 week follow-up
Time Frame: 42 Days after the End of Treatment visit
Population: Participants in the Intent to Treat Population with Global Success at End of Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 750 mg
Number analyzed (Participants) | 21
Participants | 1

5. Secondary Outcome: Percentage of Participants Surviving 42 and 84 Days
Description: Percentage of participants Surviving at Day 42 and Day 84 after Day 1 (first dose of study drug)
Time Frame: Day 42 and Day 84 after first dose of study drug
Population: Intent to Treat Population (ITT): all subjects who were enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrexafungerp 750 mg
Number analyzed (Participants) | 30
Participants
  Day 42: Survived | 24
  Day 42: Died | 4
  Day 42: Unknown survival status | 2
  Day 84: Survived | 19
  Day 84: Died | 8
  Day 84: Unknown survival status | 3

ADVERSE EVENTS:
Time Frame: From signing of Informed Consent to Week 6 follow up (up to 132 Days)
Groups:
- Ibrexafungerp 750mg: Single Arm: Oral ibrexafungerp was to be given as 750 mg BID (total daily dose = 1500 mg) on Days 1 and 2, followed by oral ibrexafungerp 750 mg QD (total daily dose = 750 mg) from Day 3 onwards for up to 90 days
Arm/Group | Ibrexafungerp 750mg
All-Cause Mortality (participants affected / at risk) | 8/30
Serious Adverse Events (participants affected / at risk) | 11/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp 750mg (N=30)
Abdominal sepsis (Infections and infestations) | 1
COVID-19 Pneumonia (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Systemic Candida (Infections and infestations) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Hematemesis (Gastrointestinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Volvulus of small bowel (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrexafungerp 750mg (N=30)
Diarrhoea (Gastrointestinal disorders) | 11
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 2
Blood potassium increased (Investigations) | 2
Escherichia test positive (Investigations) | 2
Liver function test abnormal (Investigations) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Hypernatraemia (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Candida infection (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Pneumonia klebsiella (Infections and infestations) | 2
Septic shock (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Seizure (Nervous system disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Anaemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Bradycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 2
Pyrexia (General disorders) | 3
Multiple organ dysfunction syndrome (General disorders) | 2
Pain (General disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 2
Insomnia (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03363841/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03363841/SAP_001.pdf